CLINICAL TRIAL: NCT06314438
Title: Co-Developing and Piloting Culturally-Responsive Informational Materials About Autism for Families of Young Children: Employing a Train-the-Trainer Implementation Model Within a Nonprofit Setting
Brief Title: Culturally-Responsive Curriculum for Caregivers With Children at Autism Likelihood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Hannah Benavidez, Graduate Fellow, School of Medicine: Pediatrics, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00017189; UL1TR002319 (NIH)
Record Dates: First submitted 2023-12-21; First posted 2024-03-18 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Autism; Development Delay
MeSH Terms: conditions — Autistic Disorder; Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Care Project workbook (Experimental): Caregivers will be administered the Family Care Project workbook.
  Interventions: Behavioral: Family Care Project

INTERVENTIONS:
Behavioral: Family Care Project — Caregivers will be administered the Family Care Project workbook.

SUMMARY:
The goal of this clinical trial is to examine how helpful and relevant the Family Care Project workbook is for families from culturally and linguistically diverse backgrounds who have a young child at autism likelihood. The main questions this trial aims to answer are:

* Is the Family Care Project workbook useful for families?
* Is the Family Care Project workbook easy to use?
* Can the Family Care Project be implemented by non-profit workers who do not have health backgrounds?

Participants will complete surveys that elicit their feedback on their use of the workbook.

DETAILED DESCRIPTION:
Access to early, evidence-based autism-specific treatment can profoundly improve long-term outcomes for children with Autism Spectrum Disorder (ASD). However, current estimates reveal an eight-month to three-year gap between caregiver first concerns about their child's ASD-related behaviors and receipt of ASD-specific services. This prolonged time-period between caregiver first concerns and receipt of ASD-specific services is characterized by elevated parenting stress, increased child behavioral challenges, and reduced quality of life, even compared to families of children with non-ASD developmental concerns. Unfortunately, culturally and linguistically diverse (CALD) communities experience lengthier time-periods between first concerns and receipt of services, report increased difficulty accessing timely diagnostic and treatment services, and ultimately experience worse health outcomes compared to White communities. The investigators will partner with Mother Africa, a local non-profit organization, to 1) co-design culturally-responsive caregiver-focused educational materials to support CALD families with young children who have social communication delays or ASD and 2) develop a novel route for dissemination of information and materials within non-profit organizations, which are often the preferred entry-point for accessing healthcare information and services for underserved populations, rather than traditional medical facilities. The educational materials will support caregiver and child well-being by increasing caregiver knowledge and use of ASD specific parenting strategies as well as increasing caregiver awareness and use of local ASD resources. This planned research has the potential to effect programmatic changes in the services and settings available to support CALD communities during the early years of a child's ASD condition and thereby improve child and caregiver outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Has a child who screens at likelihood on the Ages and Stages Questionnaire
* Speaks one of the following languages: Arabic, Mai Mai, Swahili, French, Tigrinya, Dari

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Stone, PhD, Principal Investigator — University of Washington
Locations (1):
- Mother Africa, Kent, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Our community organization recruit eligible families.
Pre-assignment Details: No participants were excluded from participation in this study.
Groups:
- Family Care Project Workbook-Caregivers: Caregivers will be administered the Family Care Project workbook.
- Family Care Project Workbook-nonspecialist Providers: Non-specialist providers administered the Family Care Project workbook to caregivers.
Period: Overall Study
Arm/Group | Family Care Project Workbook-Caregivers | Family Care Project Workbook-nonspecialist Providers
Started | 35 | 6
Completed | 35 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Family Care Project Workbook-nonspecialist Providers.: Nonspecialist providers will administer the Family Care Project workbook to caregivers
- Total: Total of all reporting groups
Arm/Group | Family Care Project Workbook-caregivers | Family Care Project Workbook-nonspecialist Providers. | Total
Number analyzed (Participants) | 35 | 6 | 41
Age, Categorical [Count of Participants; unit: Participants] — Demographic Survey
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 35 | 6 | 41
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic Survey
  Participants
    Female | 35 | 6 | 41
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Demographic Survey
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 35 | 6 | 41
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Demographic Survey
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 5 | 1 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 24 | 4 | 28
    White | 6 | 1 | 7
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Staff Competence in Assisting Families with Children at-autism Likelihood Survey (self-report) [Mean (Standard Deviation); unit: score on a scale] — Through a study-specific survey, staff will self-report their competence in identifying caregiver concerns, helping caregivers access services, providing new parenting strategies to caregivers, and helping caregivers set up a self-care plan. They will complete these questions via a survey and rate a score on a Likert scale of agreement with statements that reflect these topics. Higher scores indicate greater competence in assisting families with children at-autism likelihood.
  Scale title: Family Support Sister Self-Competence in Family Care Project Topics Minimum score: 1 Maximum score: 5 Population: Only includes non-specialist providers who delivered Family Care Project to caregivers.
  Caregivers did not complete this baseline measure
  score on a scale
    number analyzed (Participants) | 0 | 6 | 6
    (all) |  | 4.70 (0.47) | 4.70 (0.47)
The Maternal Self-Efficacy Scale Questionnaire [Mean (Standard Deviation); unit: score on a scale] — This questionnaire is a validated measure of caregivers' beliefs about their performance (i.e., self-efficacy) in caregiving tasks. Caregivers will fill out the survey online. They will complete these questions via a survey and rate a score on a Likert scale of agreement. Higher scores indicate greater maternal self-efficacy.
  Scale title: Maternal Self-Efficacy Scale Minimum score: 1 Maximum score: 4 Population: Only includes caregivers who completed the Family Care Project and the maternal self-efficacy survey. Does not include non-specialist providers in study. 12 caregivers did not complete the entire survey and data could not be reported for these caregivers
  score on a scale
    number analyzed (Participants) | 23 | 0 | 23
    (all) | 3.28 (0.74) |  | 3.28 (0.74)
Caregiver Knowledge and Use of Behaviors that Support Children at autism-likelihood Survey [Mean (Standard Deviation); unit: score on a scale] — Caregivers answer questions about their knowledge of child development, navigating appropriate child services, setting up a visual support, and creating a self-care plan. This survey is study-specific and created based on the curriculum topics. It will be filled out via online survey and caregivers will rate a score on a Likert scale of agreement with statements that reflect these topics. Higher scores indicate greater knowledge and use of behaviors to support children at autism-likelihood.
  Scale title: Caregiver Knowledge and Use Minimum score: 1 Maximum score: 5 Population: Includes only caregivers who completed Family Care Project and completed the survey. Non-specialist providers did not complete this measure. 15 caregivers did not complete the survey in its entirety in order to be reported.
  score on a scale
    number analyzed (Participants) | 20 | 0 | 20
    (all) | 3.81 (0.82) |  | 3.81 (0.82)
Current Services Utilized by Families to Support Children at autism-likelihood Survey [Count of Participants; unit: Participants] — Through a study-specific survey, caregivers will answer questions about their child's developmental diagnostic evaluations or current developmental services in the community. They will complete the survey online. Population: Includes only caregivers who completed the Family Care Project and survey. Non-specialist providers did not complete this survey.
  Participants
    number analyzed (Participants) | 35 | 0 | 35
    Caregivers who had received a diagnostic or intervention referral before Family Care Project | 5 |  | 5
    Caregivers who did not received a diagnostic or intervention referral before Family Care Project | 30 |  | 30

OUTCOME MEASURES:

1. Primary Outcome: Staff Training Feedback Survey of Implementation Properties (Self-report)
Description: Through a study-specific survey, staff will answer questions about the acceptability, feasibility, and appropriateness of the training. Staff will also have the opportunity to offer suggestions for improvements to the training curriculum. This questionnaire is administered online.
Time Frame: 1 week after staff complete training in Family Care Project, which is 1 week before the pilot commences
Population: It was supposed to be non-specialist providers who completed the web-based tutorial (n=6); however, data was not collected properly because there was an issue with the online questionnaire, specifically the Likert scale was presented incorrectly (i.e., the neutral and slightly agree were accidentally combined into "NeutraCompletelyee") and some providers chose this anchor. Therefore, we cannot infer what the providers intended in their selection of this inaccurate anchor.
Arm/Group | Family Care Project Workbook-caregivers | Family Care Project Workbook-nonspecialist Providers
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Staff Competence in Assisting Families With Children At-autism Likelihood Survey (Self-report)
Description: Through a study-specific survey, staff will self-report their competence in identifying caregiver concerns, helping caregivers access services, providing new parenting strategies to caregivers, and helping caregivers set up a self-care plan. They will complete these questions via a survey and rate a score on a Likert scale of agreement with statements that reflect these topics. Higher scores indicate greater competence in assisting families with children at-autism likelihood.
  Scale title: Family Support Sister Self-Competence in Family Care Project Topics Minimum score: 1 Maximum score: 5
Time Frame: 1 week after implementation of Family Care Project with pilot families
Population: All non-specialist providers who delivered Family Care Project to caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Care Project Workbook-caregivers | Family Care Project Workbook-nonspecialist Providers
Number analyzed (Participants) | 0 | 6
score on a scale |  | 4.73 (0.26)
Statistical Analysis 1: Comparison: Family Care Project Workbook-caregivers; Test type: Equivalence — paired samples t test with significance set at 0.05 p value; p = 0.34, t-test, 2 sided

3. Primary Outcome: The Maternal Self-Efficacy Scale Questionnaire
Description: This questionnaire is a validated measure of caregivers' beliefs about their performance (i.e., self-efficacy) in caregiving tasks. Caregivers will fill out the survey online. They will complete these questions via a survey and rate a score on a Likert scale of agreement. Higher scores indicate greater maternal self-efficacy.
  Scale title: Maternal Self-Efficacy Scale Minimum score: 1 Maximum score: 4
Time Frame: During the last session of the Family Care Project, which is approximately 4-6 weeks after the start of the pilot depending on family preferences
Population: Caregivers who completed the Family Care Project and the maternal self-efficacy survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Care Project Workbook-caregivers | Family Care Project Workbook-nonspecialist Providers
Number analyzed (Participants) | 23 | 0
score on a scale | 3.48 (0.51) |
Statistical Analysis 1: Comparison: Family Care Project Workbook-caregivers; Test type: Equivalence — paired samples t test with significance level at 0.05; p = 0.05, t-test, 2 sided

4. Primary Outcome: Caregiver Knowledge and Use of Behaviors That Support Children at Autism-likelihood Survey
Description: Through a study-specific survey, caregivers will answer questions about their knowledge of child development, navigating appropriate child services, setting up a visual support, and creating a self-care plan. They will also answer questions about whether they have used a visual support or implemented a self-care routine. This survey is study-specific and created based on the curriculum topics. It will be filled out via online survey and caregivers will rate a score on a Likert scale of agreement with statements that reflect these topics. Higher scores indicate greater knowledge and use of behaviors to support children at autism-likelihood.
  Scale title: Caregiver Knowledge and Use Minimum score: 1 Maximum score: 5
Time Frame: as for outcome 3
Population: Caregivers who completed Family Care Project and completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Care Project Workbook-caregivers | Family Care Project Workbook-nonspecialist Providers
Number analyzed (Participants) | 20 | 0
score on a scale | 4.46 (0.55) |
Statistical Analysis 1: Comparison: Family Care Project Workbook-caregivers; Test type: Equivalence — paired samples t test with significance set at 0.05 p value; p < 0.01, t-test, 2 sided

5. Primary Outcome: Current Services Utilized by Families to Support Children at Autism-likelihood Survey
Description: Through a study-specific survey, caregivers will answer questions about their child's developmental diagnostic evaluations or current developmental services in the community. They will complete the survey online.
Time Frame: as for outcome 3
Population: Caregivers who completed the Family Care Project and survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Family Care Project Workbook-caregivers | Family Care Project Workbook-nonspecialist Providers
Number analyzed (Participants) | 35 | 0
Participants
  Caregivers who connected with diagnostic intervention services for their child | 17 |
  Caregivers who did not get connected with local developmental or autism services | 18 |

6. Primary Outcome: Family Care Project Feedback Survey of Implementation Properties
Description: Through a study-specific survey, mother africa staff and caregivers will answer questions about the acceptability, feasibility, and appropriateness of the Family Care Project and suggestions for revisions. They will fill out questions on an online survey.
  It will be filled out via online survey and all participants will rate a score on a Likert scale of agreement with statements about the acceptability, feasibility, and/or appropriateness of the Family Care Project. Higher scores indicate greater acceptability, feasibility, and/or appropriateness of the Family Care Project.
  Scale title: Family Care Project Feedback Minimum score: 1 Maximum score: 5
Time Frame: as for outcome 3
Population: Caregivers and non-specialist providers who completed the surveys. All participated in Family Care Project (either received it or delivered it).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Care Project Workbook-caregivers | Family Care Project Workbook-nonspecialist Providers
Number analyzed (Participants) | 35 | 6
score on a scale
  Appropriateness | 4.23 (0.72) | 4.56 (0.62)
  Acceptability | 4.54 (0.60) | 4.78 (0.43)
  Feasibility: number analyzed (Participants) | 0 | 6
  Feasibility |  | 4.67 (0.49)

ADVERSE EVENTS:
Time Frame: We did not formally collect adverse event data during study.
Description: Deaths and adverse events were not assessed
Arm/Group | Family Care Project Workbook
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT06314438/Prot_SAP_000.pdf